CLINICAL TRIAL: NCT05180825
Title: A Randomized and Controlled Phase II Protocol in Non NF1 Pediatric and AYA (Adolescent and Young Adults) Patients Bearing a Newly Diagnosed Low Grade Glioma With Wild Type BRAF Gene Comparing a Daily Oral MEK Inhibitor (Trametinib) Versus Weekly Vinblastine for 18 Months
Brief Title: Pediatric Low Grade Glioma - MEKinhibitor TRIal vs Chemotherapy
Acronym: PLGG - MEKTRIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7830
Record Dates: First submitted 2021-11-25; First posted 2022-01-06 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Grade 1 Glioma; Mixed Glio-neuronal Tumors; Pleomorphic Xanthoastrocytoma
MeSH Terms: conditions — Astrocytoma | interventions — trametinib; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trametinib experimental arm (Experimental): the experimental arm will be Mekinist© (Trametinib) taken orally each day with a 18-course schedule of 4 weeks each.
  Interventions: Drug: Trametinib
- Vinblastine control arm (Active Comparator): the control arm will be the weekly intra-venous Vinblastine (Velbe©) during 18 courses of 4 weeks each
  Interventions: Drug: Vinblastine

INTERVENTIONS:
Drug: Trametinib — Mekinist© (Trametinib) taken orally each day with a 18-course schedule of 4 weeks each.
  Arms: Trametinib experimental arm
Drug: Vinblastine — weekly intra-venous Vinblastine (Velbe©) during 18 courses of 4 weeks each
  Arms: Vinblastine control arm

SUMMARY:
Pediatric low-grade glioma (PLGG) is a heterogeneous group of WHO grade I and II brain tumors, associated with a 10-year overall survival of 90%. It is the most common form of primary central nervous system (CNS) tumor arising during childhood, adolescence and young adulthood, accounting for over 30% of CNS tumors in this age group. A large group of PLGG patients will benefit from a complete resection of their tumor. Nevertheless, PLGG can occur anywhere and can be in some locations associated with neurological symptoms, unresectable or radiological progressive tumors that need medical treatments rapidly to avoid long-term sequelae. The current problem during this first line therapy is to improve tumor response, overall survival rate, as well as progression free survival. In our study, we will focus on a specific group of PLGGs without any congenital NF1 mutation and with a wild-type BRAF gene in the tumor. In this subgroup, for instance, the PFS is not increasing anymore above 50% at 3 years independently from the chemotherapeutic scheme. The two current standard therapies are carboplatin plus vincristine during 81 weeks or a weekly IV administration of vinblastine during 70 weeks. The most recent Canadian approach with vinblastine seems to have the same PFS rate, but with a better daily tolerance and less toxicities than the carboplatin/vincristine combination. Therefore, it is becoming the new standard approach in those patients. Nevertheless, we need to improve more their outcome with less recurs and a better first-line tumor response. The recent molecular discoveries involving the Ras/mitogen-activated protein kinase pathway in those PLGG is opening a new era with specific targeted therapies that might be the key to improve their survivals and giving hope to less treatment lines and a better tumor response. Therefore, we designed a prospective open randomized phase II study, named PLGG-MEKTRIC, comparing the experimental arm (a daily MEK inhibitor, Trametinib, Mekinist©) to a standard arm comprising weekly vinblastine during 18 courses of 4 weeks each. The study will enroll 134 patients with a PLGG during childhood, adolescence or young adulthood with no NF1-related disease and without any BRAFv600 mutation located in brain or spine. 67 patients, in each treatment arm, are planned to be enrolled to answer our primary objective. This primary objective will be to determine in the experimental arm a 20% superiority of the 3-year PFS rate in comparison with the standard treatment administered during 18 courses (e.g. 72 weeks). A stratification of the patients will be done in both arms based on molecular tumor results and brain/spine locations to obtain two equivalent arms to be analyzed.

The recruitment time will be 36 months and the complete follow-up of each patient will last 3 years. The secondary objectives will be in both arms: the tumor response rate at 24 and 72 weeks of treatment, the 3-year PFS and OS rates and the frequency of AE/SAE/SUSAR (Adverse Event/Serious Adverse Event) based on CTCAE criteria during the 3 years after the first administration. A Quality of Life (QoL) assessment, based on PEDsQL questionnaires, at 24 weeks, at the end of treatment and 3 years after 1st treatment administration in both arms will be part of this study. Finally, 3-year PFS and OS will be analyzed according to molecular biomarkers and visual assessment (LogMar scale) in each arm. An economic analysis is also planned as an ancillary study to determine a cost effectiveness of the best arm and complementary ancillary molecular studies are already organized. In the future, we hope to push forward this new-targeted therapy as a referenced first line treatment of pediatric PLGG to obtain the best tolerance and positive long-term impact and to extend our knowledge of MEK inhibitor impact in molecular subgroups and in optical pathway locations. We also plan to do a "switch" strategy in patients relapsing in standard arm and we will propose systematically to those patients the experimental treatment (MEK inhibitor ).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 1 month to ≤ 25 years
* Signed written informed consent prior to study participation of the legal representatives and the patient if the patient can understand the impact of clinical trial and to give consent. For patients above 18 years, their written informed consent will be obtained.
* Patient may be under guardianship or curatorship (for patient under legal guardianship, authorization is given by the legal representative of the patient under guardianship. For patient under curatorship, consent will be obtained from the adult assisted by his or her legal curator
* Histologically proven grade 1 glioma/mixed glio-neuronal tumors or pleomorphic xanthoastrocytoma (PXA) confirmed by local referee and the centrally pathology reviewing
* Determination of a negative BRAFv600 mutation by immunohistochemistry and/or molecular methods
* Systematic determination 7q34 duplication status or KIAA1549-BRAF fusion
* Midline tumors without proven histone H3 mutations
* Diffuse glioma without IDH1 mutation
* Collection of fresh frozen tumor tissues and/or paraffin-embedded samples for further molecular biomarker testing
* Sus-tentorial, optic pathway, midline and spine locations allowed
* Karnofsky or Lansky ≥ 50%
* Criteria for post-surgical treatment: severe visual or neurological symptoms at diagnosis, clinical deterioration of visual or neurological symptoms or radiological progression. The radiological progression is defined as an increase of solid part of the tumor of more than 25% compared to the pre-baseline MRI-imaging over a time period of at least 3 months or the occurrence of new metastatic lesions.
* Infants below one year of age with chiasmatic and/or hypothalamic tumor will be treated immediately after surgery, independently from neurological and/or visual evolution
* Females of child-bearing potential must be willing to practice highly effective contraception during all treatment and until 6 months after the last dose of study drugs' administration. Additionally, females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to start of study drugs. Boys with reproductive potential must be willing to use condom and consider contraception for partner women of childbearing potential during treatment and until 4 months after the last study drugs' administration.
* Patients must have adequate bone marrow function defined as: absolute neutrophil count (ANC) ≥ 1500/µL; platelets ≥ 100,000/µL and hemoglobin ≥ 9.0 g/dl
* Patients must have adequate liver function within 7 days prior to screening: bilirubin (sum of unconjugated and conjugated) ≤ 1.5 ULN for age, ALT and AST ≤ 2.5 x upper limit of normal, alkaline phosphatase ≤ 4 x upper limit of normal, INR/PTT < 1.5 x upper limit of normal,
* Patients must have adequate renal function within 7 days prior to screening: serum creatinine < 1.5 x upper limit of normal for age and a creatinine clearance > 60 ml/min for 1.73 m2
* Cardiac function defined as a corrected QT (QTcF) interval < 480 msec, LVEF ≥ lower limit of normal (LLN) by echocardiogram (ECHO)
* Adequate blood pressure control (smaller or equal to the 95th percentile for patient's age, height and gender)
* Patients are willing and able to comply with scheduled visits, treatment plan, laboratory tests and study procedures
* Guardians (in case of patients under 18 years) or patient if above 18 years must be affiliated to or a beneficiary of health insurance system.

Non-inclusion criteria

* Patients presenting a neurofibromatosis type 1 (NF1) congenital disease
* Pure optic nerve glioma, limited to one nerve and without optic chiasma infiltration.
* Completely resected tumors
* Previous treatment except tumor surgery
* Pregnancy and lactation
* Participation in other clinical trials
* Prior non-surgical therapy for this tumor
* Diffuse intrinsic pontine glioma (DIPG), even if histologically diagnosed as WHO grade II
* Subependymal giant astrocytoma (SEGA) in patients with TSC
* Patient having a known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis B or C
* Known hypersensitivity to drugs or excipients
* History of another malignancy
* History of current uncontrolled infection

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2031-11-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the 3-year PFS (Progression Free Survival rates) comparing the two arms (standard vs experimental). | At 3 years

SECONDARY OUTCOMES:
the OS rate: | At 3 years
  the OS calculation will take into account the survival measured from time of 1st treatment administration up to death
the tumor response based on the international and recognized RANO criteria, | at 24 weeks
  the analysis comparing the 2 arms will be based on overall response rate (ORR) by central independent radiological review assessment. The analysis will be conducted in all patients at least at 24 weeks of completed treatment or earlier for the patients who have discontinued for progression reasons. The tumor response will classify the patients in 2 groups: PD subgroup versus CR/PR/SD subgroup.
the tumor response based on the international and recognized RANO criteria, | at 72 weeks
  the analysis comparing the 2 arms will be based on overall response rate (ORR) by central independent radiological review assessment. The analysis will be conducted in all patients at least at 24 weeks of completed treatment or earlier for the patients who have discontinued for progression reasons. The tumor response will classify the patients in 2 groups: PD subgroup versus CR/PR/SD subgroup.
the frequency and description of AE (adverse event)/SAE (serious adverse event) | At the end of Cycle 18 (each cycle is 28 days)
  based on CTCAE criteria (using NCI-CTCAE version 5.0) focusing on visual disturbances, skin, intestinal and cardiac side effects in the experimental arm compared with the standard control arm.
the PFS and OS rates according to molecular biomarkers obtained with routinely done molecular analyses (RENOCLIP-LOC platform) and after centralized review of each tumor histology. | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Natacha ENTZ-WERLE, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (25):
- France (25):
  - Chu Amiens Picardie, Amiens
  - Chu D'Angers, Angers
  - Chu de Besancon, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Chu de Brest Morvan, Brest
  - CHU CAEN, Caen
  - Chu Dijon Bourgogne, Dijon
  - Chu Grenoble Alpes, Grenoble
  - Clcc Oscar Lambret Lille, Lille
  - Chu Limoges, Limoges
  - Centre Leon Berard, Lyon
  - APHM, Marseille
  - Chu Montpellier, Montpellier
  - Chu de Nice, Nice
  - Institut Curie, Paris
  - Chu Poitiers Chu La Miletrie, Poitiers
  - CHU de REIMS, Reims
  - Chu de Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - CHU Strasbourg - France, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Chu de Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif